CLINICAL TRIAL: NCT05402761
Title: Effects of Nurse-Guided Brief Behavioral Treatment for Insomnia on Sleep, Mood, and Cognition: Model Establishment and Application in Patients at the Recovery Phase Following Traumatic Brain Injury
Brief Title: Effects of Nurse-Guided BBTi for Improving Insomnia : in Patients at the Recovery Following Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202104039
Record Dates: First submitted 2022-04-04; First posted 2022-06-02 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Insomnia; Traumatic Brain Injury
Keywords: Insominia; BBTi; Traumatic Brain Injury
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nurse-guided BBTi group (Experimental): Participants will experience 4-week treatment period (2 in person and 2 via telephone).
  Interventions: Behavioral: Nurse-guided BBTi group
- Mobile-delivered BBTi group (Experimental): Participants will be shown how to download and use the app in their own mobile device after the baseline assessment.
  Interventions: Behavioral: Mobile-delivered BBTi group
- Sleep hygiene control group (No Intervention): Participants will receive sleep hygiene at the enrollment of the study and be required to maintain their usual lifestyle and medical treatment for 4 weeks.

INTERVENTIONS:
Behavioral: Nurse-guided BBTi group — On the arrival for the baseline appointment, participants will receive workbooks which include an outline and content of BBTi. In the end of week 1 and 3, nurse interventionist will meet participants to review their sleep diary data and negotiate their bedtime and wake-time schedule. During the weeks 2 and 4, participants will receive planned follow-up phone calls to assess their adherence and review progress and challenges.
  Arms: Nurse-guided BBTi group
Behavioral: Mobile-delivered BBTi group — They will use the app in conjunction with the standard BBTi procedures provided by the app, such as stimulus control, sleep restriction and audio-guided relaxation techniques (suggest to use before bedtime).
  Arms: Mobile-delivered BBTi group

SUMMARY:
nsomnia is a frequent complaint reported by patients with TBI, and exacerbates their ability to return to productive activity, which subsequently elevate related healthcare costs and burden. Existing literatures found that effects of CBTi, first-line therapy for insomnia, on post-traumatic insomnia is still debated, indicating that developing an alternative nonpharmacological therapy for alleviating insomnia following TBI is required. Besides, digital health is one of strategies to achieve precision health. Thus far, knowledge regarding whether mobile-delivered BBTi has non-inferiority effects as BBTi in treating insomnia is still lacking. Therefore, a RCT with a large sample size to examine the immediate and lasting effects of BBTi and mobile-delivered BBTi on insomnia, mood disturbances, and cognitive dysfunctions in patients following TBI at the recovery stage compared with the control participants.

DETAILED DESCRIPTION:
Background: Insomnia is highly prevalent in adults with traumatic brain injury (TBI), which in turn undermine their mood, cognitive functions, and quality of life. However, an effective non-pharmacological intervention for managing insomnia in this population is still lacking. Nurses, the first-line healthcare providers, should therefore seek an approach for managing post-TBI sleep. Brief behavioral treatment for insomnia (BBTi) is a new treatment direction for primary and comorbid insomnia; however, its treatment model has not been applied in people with neurological deficits such as TBI.

Purposes: To establish the BBTi treatment model among insomniacs in Taiwan, and to examine the immediate and lasting effects of nurse-guided BBTi and mobile-delivered BBTi on sleep, mood, and cognitive functions in adults with TBI. We hypothesize that people with TBI undergoing nurse-guided BBTi and mobile-delivered BBTi will experience greater alleviations in insomnia, mood disturbances, and cognitive dysfunctions in comparison with participants in the sleep hygiene control group.

Methods: This 3-year, assessor-blinded randomized controlled trial will employ a three-arm parallel-group design. A total of 228 TBI survivors with insomnia complaints will be randomly allocated to the nurse-guided BBTi, mobile-delivered BBTi, or sleep hygiene control group in a 1:1:1 ratio. For the nurse-guided BBTi group, all participants will experience 4-week-long BBTi via 2 in person and 2 telephone sessions. For the mobile-delivered BBTi, participants will use the apps in conjunction with the standard BBTi procedures provided by the functions of apps: "Sleep Aids" and "Relaxation therapy". For the sleep hygiene control group, they will receive usual care and sleep hygiene education. Measurement outcomes are sleep parameters measured by the Chinese version of Insomnia Severity Index, Chinese version of Epworth sleepiness scale, Chinese version of Pittsburgh sleep quality index, and 7-day actigraphy with a sleep diary. Secondary outcomes consist of mood and cognitive functions assessed using The Depression, Anxiety and Stress Scale - 21 Items, Ruff 2 & 7 test, Rey Auditory Verbal Learning Test, and Symbol Digit Modalities Test.

Questionnaires and actigraphy will be assessed in pretreatment, posttreatment, and the 6th and 12th months after treatment. A generalized estimating equation will be used to test research hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* have received a diagnosis of TBI at least 3 months before enrollment (TBI in chronic stage),
* yield an initial (i.e., rated in the emergency room) GCS score of 3-15 (mild to severe) and have GCS score of 15 when enrolling into the study,
* report lying awake for ≥30 min a night for ≥3 nights per week for ≥3 months,
* have post-TBI insomnia with a total score > 7 on the Chinese version of the insomnia severity scale (CISI) at screening,
* be able to communicate in Mandarin Chinese, and be able to complete cognitive tasks (having Rancho Los Amigos Levels of Cognitive Functioning scale score > 9)

Exclusion Criteria:

* include premorbid diagnoses of seizure,
* sleep disorders (e.g., sleep apnea, screened by using the STOP-Bang questionnaire with a score > 3),
* psychiatric diseases,
* substance abuse,
* alcoholism
* Shift workers and women who are pregnant, breastfeeding, or in the menopausal transition

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Insomnia Severity | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  The ISI consists of seven items, and each item can be rated from 0 to 4, resulting in total score ranging from 0 to 28, with higher scores indicating greater insomnia severity. A cutoff score of > 7 is used to diagnose subthreshold insomnia.
Changes in Sleep quality | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  Sleep quality will be measured by Pittsburgh Sleep Quality Index (PSQI). PSQI has 18 questions to evaluate sleep condition. The score range from 0-21, if score>5 is associated with poor sleep. The higher score means poorer sleep quality.
Changes in Daytime Sleepiness | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  Daytime Sleepiness will be measured by Epworth Sleepiness Scale (ESS). ESS has 8 questions to evaluate the condition of dozing off or falling asleep. The score range from 0-24, if score>10 is associated with daytime sleepiness.
Changes in Sleep parameters from sleep logs: sleep onset latency(SOL) | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  Sleep onset latency(SOL) is the time of duration from lying on bed to fall asleep. SOL shorter than 30 minutes is one of criteria of good sleep condition.
Changes in Sleep parameters from sleep logs: after sleep onset(WASO) | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  Wake after sleep onset(WASO) is the total time of wakefulness after sleep onset. WASO less than 30 minutes is one of criteria of good sleep condition.
Changes in Sleep parameters from sleep logs: total sleep time(TST) | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  Total sleep time(TST) is the total time of falling asleep. TST will be used to calculate sleep efficiency(SE).
Changes in Sleep parameters from sleep logs: sleep efficiency(SE) | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  Sleep efficiency(SE) is the percentage of total sleep time to time in bed. A good sleep condition should meet the criteria of SE greater than 85%.

SECONDARY OUTCOMES:
Changes in Depression | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  Depression will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of depression. The total score should be multiplied by 2 range from 0-42, if score>9 is associated with depression. The higher score means more severe depression.
Changes in Anxiety | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  Anxiety will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of anxiety. The total score should be multiplied by 2 range from 0-42, if score>7 is associated with anxiety. The higher score means more severe anxiety.
Changes in Stress | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  Stress will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of stress. The total score should be multiplied by 2 range from 0-42, if score>14 is associated with anxiety. The higher score means more severe stress.
Changes in Ruff 2 and 7 | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  The Ruff 2 & 7 test will be used to test sustained and selective aspects of visual attention. It consists of 20 trials (10 Automatic Detection trials and 10 Controlled Search trials), with three line per trial, administered consecutively in 15-s intervals, working from left to right. The Automatic Detection and Controlled Search scores will used to assess selective attention. Sustained attention is measured primarily by the Total Speed (number of correctly identified targets during the allotted 5-min duration), and Total Accuracy (number of targets identified during the 5-min duration divided by the number of possible targets) scores.
Changes in Rey Auditory Verbal Learning Test (RAVLT) | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  The RAVLT is a measure of verbal memory in which a subject is read a list of 15 words and asked to recall them after the examiner finishes reading the list. The subjects are exposed to the second list once, after which they must recall as many words as they can from the first list. After a 30-minute delay, the subjects are again asked to recall the words from the first list; they subsequently participate in a recognition trial in which they determine whether the word heard was in the first list.
Changes in Symbol digital modalities | at baseline and the 5th week and the 12th week after intervention finished and the 24th week after intervention finished
  The SDMT is a brief test of information processing speed that has become the most commonly used cognitive measure in patients with TBI. It consists of a sheet of paper with a sequence of nine symbols and nine corresponding numbers at the top. Responses can be written or oral, and for either response mode, the administration time is 5 min. A higher score indicates a more favorable performance.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Medical University, Taipei
  - Skin Kong International Health Center, Taipei